CLINICAL TRIAL: NCT05135806
Title: Feasibility Study on Remote Cognitive Assessment With Older People. A Counter-balanced Crossover Trial.
Brief Title: Remote Testing in Abbiategrasso (RTA)
Acronym: RTA
Status: Completed | Type: Observational
Sponsor: Fondazione Golgi Cenci (Other)
Responsible Party: Principal Investigator, Antonio Guaita, MD, MD, Fondazione Golgi Cenci
Other Study IDs: 03
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Assessment
Keywords: remote neuropsychological assessment; feasibility study; counterbalanced cross-over design

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Remote evaluation first: participants will undergo a comprehensive neuropsychological assessment administered remotely via telephone calls or videoconferencing. Each participant will take part to the second evaluation (face-to-face) 8 weeks later.
- Group 2: Face-to-face evaluation first: participants will undergo a comprehensive neuropsychological assessment administered face-to-face. Each participant will take part to the second evaluation (remotely via telephone calls or videoconferencing) 8 weeks later.

SUMMARY:
The remote cognitive assessment has the advantage of reaching people despite the restrictions due to the pandemic, so it is of fundamental importance both in the treatment of dementia and the research context. The scientific literature on the feasibility, acceptability and validity of remote neuropsychological assessment provides promising indications. However, the limitations related to access and familiarity with technologies in elderly populations, and to methodological aspects (e.g. the not-controlled environment, the validity of the remote assessment compared to the in-person assessment) remain to be clarified. For the present observational feasibility study, 58 older adults (65-85 years), randomly extracted among 93 eligible participants, will be recruited among donors of our Brain Bank. Participants will undergo both face-to-face and remote testing (via phone calls or videoconferencing) sessions in a counterbalanced cross-over design. The study will target (1) the recruitment rate in a study on remote testing, (2) the acceptability of remote cognitive tests and the procedures for delivering remote testing, (3) the comparability between remote and face-to-face performances on neuropsychological tests.

DETAILED DESCRIPTION:
In February and March 2021, the 237 donors of our Brain Bank, aged between 65 and 98 and living at home, were interviewed by telephone. The purpose of the survey was to collect information on how they were experiencing the isolation linked to the pandemic in the last year, on health conditions and sleep, daily habits (nutrition, movement, leisure), use of the Internet and social networks as a way to maintain contact with one's family-friend network and experiences of loneliness (Rolandi et al, 2020). In this context, the willingness to participate in a study on remote cognitive assessment by phone, personal computer or tablet was explored.

The sample size was calculated to estimate differences between testing conditions, i.e. face-to-face and remote testing (telephone or videoconference). A sample size of 52 is required to detect an effect size of 0.40 at 0.80% of power, in a paired-sample test with a normal distribution. We planned an increase in sample size of 6 participants, because the expected drop-out rate is 10% due to possible acute clinical conditions interfering with the participation in the study, or death.

For the present observational feasibility study, 58 older adults (65-85 years), randomly extracted among 93 eligible participants, will be recruited among donors of the Brain Bank who previously have expressed the willingness to adhere to the study. Participants will undergo both face-to-face and remote testing sessions in a counterbalanced cross-over design. Each individual will undergo a comprehensive neuropsychological assessment consisting of a set of cognitive tests (memory, attention, etc) administered remotely via telephone calls or videoconferencing and face-to-face. Participants will be randomly allocated to one of the two conditions (remote first or face-to-face first). Each participant will take part to the second evaluation (remote or face-to-face) 8 weeks later. To reduce learning effect bias and intra-rate variability, this procedure will be counterbalanced so that half of the participants first experience the face-to-face interaction and the other half will initially receive the videoconference administration.

ELIGIBILITY:
Inclusion Criteria:

* willingness to adhere to the study
* age between 65 and 85
* normal cognition

Exclusion Criteria:

* dementia, psychiatric or neurological diagnosis
* presence of a memory disorder with impact on the daily life reported by the person or detected by the interviewer
* previously scheduled follow-up of the Brain Bank

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: In February and March 2021, the 237 donors of the Abbiategrasso Brain Bank, aged between 65 and 98 and living at home, were interviewed by telephone. The purpose of the survey was to collect information on how they were experiencing the isolation linked to the pandemic in the last year (Rolandi et al, 2020). In this context, the willingness to participate in a study on remote cognitive assessment by phone, personal computer or tablet was explored. For the present observational feasibility study, 58 older adults (65-85 years), randomly extracted among 93 eligible participants, will be recruited among donors of the Abbiategrasso Brain Bank who previously have expressed the willingness to adhere to the study.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Day 0
  The primary outcome is the recruitment of the 58 Brain Bank donors in our study on remote cognitive assessment. Fifteen days after the informed consent is sent, the healthcare assistant will conduct telephone calls to receive confirmation of participation in a remote cognitive assessment study from the donors who previously had expressed their willingness to adhere. The healthcare assistant will collect information about the reason of refusal if any (i.e. not interested, health problems, away from home for holidays). It will also asked confirmation of the modality preferred for the remote assessment, i.e. by phone, tablet or computer.

SECONDARY OUTCOMES:
Acceptability of remote cognitive tests among aged individuals (+65 years). | Day 1 and Month 2
  Immediately following each session of cognitive evaluation (both remotely and face-to-face) participants completed an acceptability questionnaire previously developed to evaluate the response to computerised cognitive tasks in both the clinic-based and home-based setting. Participants will be required to rate the enjoyability, level of anxiety, engagement, duration and repeatability of the tasks, rating them on a five-point Likert scale: 1, not at all; 2, a little bit; 3, neutral; 4, slightly; 5, very much. The questionnaire comprises the following questions: Did the test make you anxious? Did you enjoy the test? Did you find the test interesting? Would you be happy to repeat the test? What did you think about the duration of the test?

OTHER OUTCOMES:
Comparison between remote and face-to-face performances on the Montreal Cognitive Assessment (MoCA) Audiovisual | Day 1 and Month 2
  The MoCA Audiovisual is the version of the MoCA test used for video administration with little adaptation. It is a screening test including 5-word learning (attention), animal semantic fluency (language, executive function), 6-item orientation, and delayed recall (memory). The visual section (trail making, clock drawing and the cube copy) is displayed on the video using the share screen option (range 0-30).
Comparison between remote and face-to-face performances on the MoCA 5-minute | Day 1 and Month 2
  The MoCA 5-minute is a brief version of the MoCA test with the visual elements removed and suitable for telephone administration. It is a screening test including 5-word learning (attention), animal semantic fluency (language, executive function), 6-item orientation, and delayed recall (memory). The MoCA 5-minute has been translated in Italian and it is commonly used in clinical setting (range 0-15).
Comparison between remote and face-to-face performances on the Rey Auditory Verbal Learning Test (RAVLT) | Day 1 and Month 2
  The RAVLT evaluates verbal learning and memory in young and older adults. It is designed as a list-learning paradigm in which the subject hears a list of 15 nouns and is asked to recall as many words from the list as possible. After a 15 minutes delay (performing interference non-verbal tasks), the participant is immediately asked to recall the words from the list. The RAVLT provides immediate (sum of words recalled on the 5 learning trials; range 0-75) and delayed recall scores (sum of the words recalled after 15 min; range 0-15), with higher scores indicating better performance on verbal learning and long-term memory.
Comparison between remote and face-to-face performances on the Digit span forward and backward | Day 1 and Month 2
  Digit span forward and backward are two subtests of the Wechsler Adult Intelligence Scale, assessing short-term memory and working memory respectively. Participants are asked to repeat sequences of numbers of increasing length in straight order (Digit span forward) or reverse order (Digit span backward). Performances are reported as span scores (the maximum number of digits correctly produced forwards or backwards by the subjects) (range 0-9), with higher scores indicative of better performance on short-term memory and working memory.
Comparison between remote and face-to-face performances on the alternate phonemic/semantic fluency test | Day 1 and Month 2
  The alternate phonemic/semantic fluency test measures spontaneous verbal production, executive function, processing speed and memory. It consists of three subtests: letter-cued (phonemic) fluency, category-cued (semantic) fluency and alternate phonemic/semantic fluency. The subtests are administered in the following order: phonemic, semantic and alternate fluency. In the first, the subject is asked to produce words beginning with a specified letter (F, A and S). In the second, one is asked to produced words belonging to a specified category (colours, animals and fruits). The score is obtained by the sum of the correct responses (range 0-…) within 60 seconds, with higher scores indicating better performances. In the third, the subjects have to alternate letter-cued words with category-cued words as follows: trial (1) letter A and Colours; trial (2) letter F and Animals; trial (3) letter S and Fruits. Three trials are given, each lasting 60 seconds.
Comparison between remote and face-to-face performances on the Verbal reasoning test | Day 1 and Month 2
  Verbal reasoning test evaluates the individual's ability to reason, i.e. solve problems, draw inferences and classify, based on previous knowledge.The test consists of four subtests: differences (for instance: what is the difference between glass and plate?), proverbs (for instance: what is the meaning of "The dress does not make the priest"?), nonsense (what's wrong or what's wrong with the following story?) and classifications (for instance: please, state the likeness between Milan, Rome, Naples and Venice). The score of items is attributed on the basis of predefined criteria, so that subtest scores varies between 0 and 15 (total range score 0-60), with higher scores indicative of better performance on verbal reasoning.
Comparison between remote and face-to-face performances on the Constructional praxis | Day 1 and Month 2
  Copy figure tasks are generally included in most of the common screening tests and battery administered remotely, although the high level of variability between studies. The Constructional praxis test cannot be administered by telephone, but can be drawn during the videoconference and displayed in front of the camera. Subjects are requested to copy images representing bi-dimensional and three-dimensional shape (range 0-16), with higher scores indicative of better performance on constructional ability.
Comparison between remote and face-to-face performances on the Reading the Mind in the Eyes Test (RME) | Day 1 and Month 2
  The term Theory of Mind (ToM) refers to the abilities to attribute mental states to others and to predict, describe, and explain behaviour on the basis of such mental state. ToM abilities are involved in social functioning and are affected in neurodegenerative diseases. The RME evaluates the cognitive component of ToM in adult and older people. The test consists of 36 black and white photographs depicting the eye region of adults, young and old people of both sexes. The subject is asked to indicate the term among four adjectives placed under the photograph, best describing the emotion expressed in the image (range 0-36). To limit the effect of the linguistic competences, a glossary is available to the subjects including definitions and clarifications for each of the words associated with the photos. To adapt the administration to the remote modality, the images will be projected on the shared screen.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Vaccaro, MSc, Principal Investigator — Fondazione Golgi Cenci
Locations (1):
- Golgi cenci Foundation, Abbiategrasso, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The data may be made available to third parties as aggregated data.

REFERENCES:
- [Background] Orsini, A., & Pezzuti, L. (2013). WAIS-IV. Contributo alla taratura italiana. (Giunti OS.). Firenze.
- [Background] Rolandi E, Vaccaro R, Abbondanza S, Casanova G, Pettinato L, Colombo M, Guaita A. Loneliness and Social Engagement in Older Adults Based in Lombardy during the COVID-19 Lockdown: The Long-Term Effects of a Course on Social Networking Sites Use. Int J Environ Res Public Health. 2020 Oct 28;17(21):7912. doi: 10.3390/ijerph17217912. PMID 33126634
- [Background] Backx R, Skirrow C, Dente P, Barnett JH, Cormack FK. Comparing Web-Based and Lab-Based Cognitive Assessment Using the Cambridge Neuropsychological Test Automated Battery: A Within-Subjects Counterbalanced Study. J Med Internet Res. 2020 Aug 4;22(8):e16792. doi: 10.2196/16792. PMID 32749999
- [Background] Wong A, Nyenhuis D, Black SE, Law LS, Lo ES, Kwan PW, Au L, Chan AY, Wong LK, Nasreddine Z, Mok V. Montreal Cognitive Assessment 5-minute protocol is a brief, valid, reliable, and feasible cognitive screen for telephone administration. Stroke. 2015 Apr;46(4):1059-64. doi: 10.1161/STROKEAHA.114.007253. Epub 2015 Feb 19. PMID 25700290
- [Background] DeYoung N, Shenal BV. The reliability of the Montreal Cognitive Assessment using telehealth in a rural setting with veterans. J Telemed Telecare. 2019 May;25(4):197-203. doi: 10.1177/1357633X17752030. Epub 2018 Jan 10. PMID 29320916
- [Background] Santangelo G, Siciliano M, Pedone R, Vitale C, Falco F, Bisogno R, Siano P, Barone P, Grossi D, Santangelo F, Trojano L. Normative data for the Montreal Cognitive Assessment in an Italian population sample. Neurol Sci. 2015 Apr;36(4):585-91. doi: 10.1007/s10072-014-1995-y. Epub 2014 Nov 8. PMID 25380622
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] [Italian standardization and classification of Neuropsychological tests. The Italian Group on the Neuropsychological Study of Aging]. Ital J Neurol Sci. 1987 Dec;Suppl 8:1-120. No abstract available. Italian. PMID 3330072
- [Background] Novelli, G., Papagno, C., Capitani, E., Laiacona, M., Vallar, G., & Cappa, S. (1986). Tre test clinici di ricerca e produzione lessicale: taratura su soggetti normali. Archivio Di Psicologia Neurologia e Psichiatria, (4), 477-506.
- [Background] Costa A, Bagoj E, Monaco M, Zabberoni S, De Rosa S, Papantonio AM, Mundi C, Caltagirone C, Carlesimo GA. Standardization and normative data obtained in the Italian population for a new verbal fluency instrument, the phonemic/semantic alternate fluency test. Neurol Sci. 2014 Mar;35(3):365-72. doi: 10.1007/s10072-013-1520-8. Epub 2013 Aug 21. PMID 23963806
- [Background] Serafin, M., & Surian, L. (2004). Il Test degli Occhi: uno strumento per valutare la "teoria della mente." Giornale Italiano Di Psicologia, 31(4), 839-862.
- [Derived] Vaccaro R, Aglieri V, Rossi M, Pettinato L, Ceretti A, Colombo M, Guaita A, Rolandi E. Remote testing in Abbiategrasso (RTA): results from a counterbalanced cross-over study on direct-to-home neuropsychology with older adults. Aging Clin Exp Res. 2023 Mar;35(3):699-710. doi: 10.1007/s40520-023-02343-9. Epub 2023 Jan 30. PMID 36710319